CLINICAL TRIAL: NCT04033991
Title: A Real World Retrospective Database Study of Patients Diagnosed With Metastatic and/or Advanced Renal Cell Carcinoma and Treated With Sunitinib and/or Axitinib in a Specialist United Kingdom Oncology Centre
Brief Title: Study of Patients With Metastatic and/or Advanced Renal Cell Carcinoma, Treated With Sunitinib/Axitinib.
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: X9001180
Record Dates: First submitted 2019-07-10; First posted 2019-07-26 (Actual); Results first posted 2022-02-18 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-01

CONDITIONS: Carcinoma; Renal Cell
Keywords: Carcinoma;; renal cell;; cancer;; kidney;; sunitinib;; axitinib
MeSH Terms: conditions — Carcinoma; Neoplasms | interventions — Sunitinib; Axitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with advanced RCC: Patients with a diagnosis of kidney cancer (renal cell carcinoma, advanced or metastatic)
  Interventions: Drug: Sunitinib; Drug: Axitinib

INTERVENTIONS:
Drug: Sunitinib — Tyrosine kinase inhibitor, licensed for use in treatment of renal cell carcinoma.
  Other Names: Sutent
Drug: Axitinib — Tyrosine kinase inhibitor, licensed for use in treatment of renal cell carcinoma.
  Other Names: Inlyta

SUMMARY:
Research Questions:

To understand the clinical outcomes of patients treated with sunitinib in first line and axitinib in second line in a real world setting as therapies for metastatic and/or advanced renal cell carcinoma (mRCC).

Primary Objective:

1. What is the progression free survival (PFS) of patients treated in first line with sunitinib, and stratified by Memorial Sloan-Kettering Cancer Center / International Metastatic Renal Cell Carcinoma Database Consortium (MSKCC/IMDC) risk category (favourable, intermediate, poor)?
2. What is the progression free survival (PFS) of patients treated in second line with axitinib, and stratified by MSKCC/IMDC risk category (favourable, intermediate, poor)?

DETAILED DESCRIPTION:
Research Questions:

To understand the clinical outcomes of patients treated with sunitinib in first line and axitinib in second line in a real world setting as therapies for metastatic and/or advanced renal cell carcinoma (mRCC).

Primary Objective:

1. What is the progression free survival (PFS) of patients treated in first line with sunitinib, and stratified by Memorial Sloan-Kettering Cancer Center / International Metastatic Renal Cell Carcinoma Database Consortium (MSKCC/IMDC) risk category (favourable, intermediate, poor)?
2. What is the progression free survival (PFS) of patients treated in second line with axitinib, and stratified by MSKCC/IMDC risk category (favourable, intermediate, poor)?

Secondary Objectives:

First Line:

1. What is the overall survival (OS) of all patients in first line with sunitinib, and stratified by MSKCC risk (favourable, intermediate, poor)?
2. What is the duration of therapy with sunitinib in first line (using time to treatment discontinuation [TTD]) for all patients and stratified by MSKCC risk (favourable, intermediate, poor)
3. Objective response rate (ORR)
4. Duration of objective response (complete response [CR] or partial response [PR])
5. Examine factors that predict TTD, e.g. risk stratification, or individual/grouped parameters that comprise the prognostic classification systems

   1. Less than one year from time of diagnosis
   2. Karnovsky performance status less than 80%
   3. Haemoglobin less than the lower limit of normal (e.g. less than 12 g/dl)
   4. Serum calcium great than the upper limit of normal (e.g. 10 mg/dl or : 2.5 mmol/l)
   5. Neutrophil greater than the upper limit of normal (e.g. greater than 7.0 x109 dl)
   6. Platelets greater than the upper limit of normal (e.g. greater than 400 000)
   7. Lactate dehydrogenase greater than 1.5 times the upper limit of normal
   8. Fuhrmann grade of tumour
   9. Tumour subtype e.g. clear cell versus. non-clear cell
6. Safety and tolerability data reporting for first line sunitinib

Second line:

1. What is the OS of all patients in second line with axitinib, and stratified by MSKCC risk (favourable, intermediate, poor)?
2. What is the duration of therapy with axitinib in second line (using TTD) for all patients and stratified by MSKCC risk (favourable, intermediate, poor)
3. ORR
4. Duration of objective response (CR or PR)
5. Examine factors that predict duration of TTD, e.g. risk stratification, or individual/grouped parameters that comprise the prognostic classification systems

   1. Less than one year from time of diagnosis
   2. Karnovsky performance status less than 80%
   3. Haemoglobin less than the lower limit of normal (e.g. less than 12 g/dl)
   4. Serum calcium great than the upper limit of normal (e.g. 10 mg/dl or : 2.5 mmol/l)
   5. Neutrophil greater than the upper limit of normal (e.g. greater than 7.0 x109 dl)
   6. Platelets greater than the upper limit of normal (e.g. greater than 400 000)
   7. Lactate dehydrogenase greater than 1.5 times the upper limit of normal
   8. Fuhrmann grade of tumour
   9. Tumour subtype e.g. clear cell vs. non-clear cell
6. Safety and tolerability reporting for second line axitinib

The objectives listed below will also be assessed as exploratory analyses for various patient subgroups of interest, and will be conducted if sufficient numbers of patients are available:

1. Axitinib PFS and OS, as a second line therapy following sunitinib, pazopanib, or following other Tyrosine kinase inhibitors (e.g. sorafenib)
2. Axitinib PFS and OS as a third line therapy
3. Axitinib PFS and OS post-immunotherapy (IO), taking into consideration 2nd and 3rd therapy lines, following all IO therapy options, E.g. atezolizumab/bevacizumab, nivolumab/ipilumimab, nivolumab, interleukin-2
4. For the post-sunitinib axitinib cohort: What was the duration of sunitinib therapy before patients transitioned to axitinib?
5. For the post-pazopanib axitinib cohort: What was the duration of sunitinib therapy before patients transitioned to axitinib?
6. Is the duration of therapy on first line sunitinib and/or pazopanib related to duration of therapy for second line axitinib?

ELIGIBILITY:
Inclusion criteria

1. Over the age of 18 years
2. Diagnosis of renal cell carcinoma
3. Treatment with sunitinib and/or axitinib
4. Timeframe: from database inception date (2002) until June 30, 2018.

Exclusion criteria

Patients meeting any of the following criteria will not be included in the study:

1. Under the age of 18 years
2. Diagnosis other than renal cell carcinoma
3. No treatment with sunitinib and/or axitinib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Over the age of 18 years
  2. Diagnosis of renal cell carcinoma
  3. Treatment with sunitinib and/or axitinib
  4. Timeframe: from database inception date (2002) until June 30, 2018.
Sampling Method: Non-Probability Sample
Enrollment: 684 (Actual)
Dates: Start 2019-09-27 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2020-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer UK, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Waddell T, Pillai M, Armitage K, Graham DM, Moran M, Dilleen M, Holmes S, Sleszynska-Dopiera E, Hawkins R. Real-world effectiveness of first- and second-line anti-angiogenesis therapy in RCC: analysis of a UK-based population. Future Oncol. 2024;20(33):2547-2558. doi: 10.1080/14796694.2024.2385882. Epub 2024 Oct 9. PMID 39382446
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=X9001180

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data of participants treated with first-line sunitinib and/or second-line axitinib in real world settings for metastatic renal cell carcinoma (mRCC) and/or advanced renal cell carcinoma (aRCC), from 2002 until 30 June 2018, were retrieved from Christie National Health Service (NHS) database. Available data were extracted, curated and analyzed during approximately 1.2 years of this retrospective, observational study.
Groups:
- Participants With mRCC and/or aRCC: Participants who met the selection criteria, diagnosed with mRCC and/or aRCC, received sunitinib as first-line treatment and/or axitinib as second-line treatment from 2002 till 30 June 2018, according to normal routine healthcare practice in real-world setting, were included in this study. Data of these participants were derived from Christie NHS database.
Period: Overall Study
Arm/Group | Participants With mRCC and/or aRCC
Started | 684
Participants Who Took First-line Sunitinib Therapy | 622
Participants Who Took Second-line Axitinib Therapy | 121
Participants Who Took First-line Sunitinib Therapy and Then Second-line Axitinib Therapy | 59
Participants Who Took Drugs Other Than Sunitinib as First-line and Then Second-line Axitinib Therapy | 62
Completed | 684
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all eligible participants with mRCC and/or aRCC, received sunitinib as first-line treatment and/or axitinib as second-line treatment from 2002 till 30 June 2018.
Arm/Group | Participants With mRCC and/or aRCC
Number analyzed (Participants) | 684
Age, Customized [Count of Participants; unit: Participants]
  Less than (<) 65 years | 301
  Greater than or equal to (>=) 65 to <75 years | 247
  >=75 to <84 years | 124
  Greater than or equal to (>=) 85 years | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 234
  Male | 450
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS was duration measured from the first date of each treatment line to the date of disease progression (PD), end of treatment date or date of death. Participants who were on treatment were censored on 30 June 2018. If a participant stopped due to toxicity, the earliest date from the date of progression or end of treatment date was assigned. PD per Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1 was defined as at least a 20 percent (%) increase in sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 millimeter (mm). The appearance of one or more new lesions was also considered progression.
Time Frame: From start of treatment to PD, death or end of treatment, whichever occurred first, from inception of database (2002) until 30 June 2018, anytime in these 16 years (from the data retrieved and observed retrospectively for approximately 1.2 years)
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Participants With mRCC and/or aRCC: First Line Sunitinib Treatment: Participants who met the selection criteria, diagnosed with mRCC and/or aRCC, received sunitinib as first-line treatment from 2002 till 30 June 2018, according to normal routine healthcare practice in real-world setting, were included in this reporting arm. Data of these participants were derived from Christie NHS database.
- Participants With mRCC and/or aRCC: Second Line Axitinib Treatment: Participants who met the selection criteria, diagnosed with mRCC and/or aRCC, received axitinib as second-line treatment from 2002 till 30 June 2018, according to normal routine healthcare practice in real-world setting, were included in this reporting arm. Data of these participants were derived from Christie NHS database.
Arm/Group | Participants With mRCC and/or aRCC: First Line Sunitinib Treatment | Participants With mRCC and/or aRCC: Second Line Axitinib Treatment
Number analyzed (Participants) | 622 | 121
Months | 8.394 [7.556 to 9.889] | 6.177 [4.928 to 9.331]

2. Primary Outcome: Progression Free Survival (PFS): Memorial Sloan-Kettering Cancer Center (MSKCC) Stratification
Description: PFS: first date of each treatment line to the date of PD, end of treatment date or date of death. Participants who were on treatment were censored on 30 June 2018. If a participant stopped due to toxicity, the earliest date from date of PD or end of treatment date was assigned. MSKCC criteria had 5 risk factors: Karnofsky performance status (KPS) <80% (ability to perform ordinary tasks, 0 [dead] -100 [normal]); time from diagnosis to start of systemic therapy <12 months; hemoglobin <lower limit of normal (LLN); lactate dehydrogenase 1.5*upper limit of normal (ULN); corrected serum calcium >10 milligram per deciliter (mg/dL). Present risk factors were added, and participants were stratified as: favorable (0 factor), intermediate (1-2 factors), poor (>=3 factors). PD: >=20% increase in sum of diameters of target lesions, taking as reference smallest sum on study, the sum must also demonstrate an absolute increase of at least 5 mm. Appearance of 1 or more new lesions was considered PD.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants with mRCC and/or aRCC, received sunitinib as first-line treatment and/or axitinib as second-line treatment from 2002 till 30 June 2018. Here "Number Analyzed" signifies number of participants evaluable for specified rows.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Participants With mRCC and/or aRCC: First Line Sunitinib Treatment | Participants With mRCC and/or aRCC: Second Line Axitinib Treatment
Number analyzed (Participants) | 622 | 121
Months
  Favorable: number analyzed (Participants) | 122 | 19
  Favorable | 14.784 [11.729 to 20.008] | 12.649 [4.895 to 15.639]
  Intermediate: number analyzed (Participants) | 378 | 72
  Intermediate | 8.986 [7.589 to 10.021] | 8.903 [5.290 to 11.762]
  Poor: number analyzed (Participants) | 85 | 17
  Poor | 2.628 [1.774 to 4.600] | 1.610 [0.460 to 2.661]
  Unknown/missing (no information available): number analyzed (Participants) | 37 | 13
  Unknown/missing (no information available) | NA [NA to NA] — Median and 95% confidence interval (CI) was not calculated as no information was available for these participants. | NA [NA to NA] — Median and 95% CI was not calculated as no information was available for these participants.
Statistical Analysis 1: Comparison: Participants With mRCC and/or aRCC: First Line Sunitinib Treatment; Data were compared statistically across all 3 categories (favorable, intermediate and poor); Test type: Other; p < 0.0001, Log Rank
Statistical Analysis 2: Comparison: Participants With mRCC and/or aRCC: Second Line Axitinib Treatment; Data were compared statistically across all 3 categories (favorable, intermediate and poor); Test type: Other; p < 0.0001, Log Rank

3. Primary Outcome: Progression Free Survival (PFS): International Metastatic Renal Cell Carcinoma Database Consortium (IMDC) Stratification
Description: PFS: duration measured from first date of each treatment line to the date of PD, end of treatment date or date of death. Participants who were on treatment were censored on 30 June 2018. If a participant stopped due to toxicity, the earliest date from date of PD or end of treatment date was assigned. IMDC criteria had 6 risk factors: KPS <80% (ability to perform ordinary tasks, 0 [dead] -100 [normal]); time from diagnosis to start of systemic therapy <12 months; corrected serum calcium >10 mg/dL; neutrophils and platelets >LLN; hemoglobin <LLN. Present risk factors were added, and then participants were stratified as: favorable (0 factor), intermediate (1-2 factors), poor (>=3 factors). PD: >=20% increase in sum of diameters of target lesions, taking as reference smallest sum on study, the sum must also demonstrate an absolute increase of at least 5 mm. Appearance of 1 or more new lesions was also considered PD.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Participants With mRCC and/or aRCC: First Line Sunitinib Treatment | Participants With mRCC and/or aRCC: Second Line Axitinib Treatment
Number analyzed (Participants) | 622 | 121
Months
  Favorable: number analyzed (Participants) | 108 | 21
  Favorable | 13.979 [10.382 to 18.497] | 12.649 [5.749 to 15.639]
  Intermediate: number analyzed (Participants) | 308 | 65
  Intermediate | 9.955 [8.082 to 12.156] | 7.162 [5.158 to 10.842]
  Poor: number analyzed (Participants) | 184 | 31
  Poor | 5.569 [4.830 to 6.275] | 2.990 [1.708 to 5.651]
  Unknown/missing (no information available): number analyzed (Participants) | 22 | 4
  Unknown/missing (no information available) | NA [NA to NA] — Median and 95% CI was not calculated as no information was available for these participants. | NA [NA to NA] — Median and 95% CI was not calculated as no information was available for these participants.
Statistical Analysis 1: Comparison: Participants With mRCC and/or aRCC: First Line Sunitinib Treatment; Data were compared statistically across all 3 categories (favorable, intermediate and poor); Test type: Other; p < 0.0001, Log Rank
Statistical Analysis 2: Comparison: Participants With mRCC and/or aRCC: Second Line Axitinib Treatment; Data were compared statistically across all 3 categories (favorable, intermediate and poor); Test type: Other; p = 0.0068, Log Rank

4. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time between the index date and the date of death from any cause. Participants who were still alive at the study end date or the last visit date available were censored. Index date: date of initiation of first-line sunitinib therapy and second-line axitinib therapy.
Time Frame: From index date until death, from inception of database (2002) until 30 June 2018, anytime in these 16 years (from the data retrieved and observed retrospectively for approximately 1.2 years)
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Participants With mRCC and/or aRCC: First Line Sunitinib Treatment | Participants With mRCC and/or aRCC: Second Line Axitinib Treatment
Number analyzed (Participants) | 622 | 121
Months | 18.333 [15.770 to 20.435] | 15.836 [12.025 to 20.370]

5. Secondary Outcome: Overall Survival (OS): Memorial Sloan-Kettering Cancer Center (MSKCC) Stratification
Description: OS was defined as the time between the index date and the date of death from any cause. Participants who were still alive at the study end date or the last visit date available were censored. MSKCC criteria had 5 risk factors: KPS <80% (ability to perform ordinary tasks, 0 [dead] -100 [normal]); time from diagnosis to start of systemic therapy <12 months; hemoglobin <LLN; lactate dehydrogenase 1.5* ULN; corrected serum calcium >10.0 mg/dL. Present risk factors were added, and then participants were stratified in following prognosis group: favorable (0 factor), intermediate (1-2 factors), poor (>=3 factors), unknown/missing = no information available. Index date: date of initiation of first-line sunitinib therapy and second-line axitinib therapy.
Time Frame: as for outcome 4
Population: Analysis population included all eligible participants with mRCC and/or aRCC, received sunitinib as first-line treatment and/or axitinib as second-line treatment from 2002 till 30 June 2018. Here, "Number Analyzed" signifies number of participants evaluable for specified rows.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Participants With mRCC and/or aRCC: First Line Sunitinib Treatment | Participants With mRCC and/or aRCC: Second Line Axitinib Treatment
Number analyzed (Participants) | 622 | 121
Months
  Favorable: number analyzed (Participants) | 122 | 19
  Favorable | 40.246 [30.357 to 47.540] | NA [NA to NA] — Median and 95% CI was not estimable due to low number of participants with events.
  Intermediate: number analyzed (Participants) | 378 | 72
  Intermediate | 18.497 [15.934 to 20.468] | 16.164 [11.630 to 20.370]
  Poor: number analyzed (Participants) | 85 | 17
  Poor | 5.322 [3.614 to 6.998] | 2.694 [1.840 to 8.444]
  Unknown/missing (no information available): number analyzed (Participants) | 37 | 13
  Unknown/missing (no information available) | NA [NA to NA] — Median and 95% CI was not calculated as no information was available for these participants. | NA [NA to NA] — Median and 95% CI was not calculated as no information was available for these participants.
Statistical Analysis 1: Comparison: Participants With mRCC and/or aRCC: First Line Sunitinib Treatment; Data were compared statistically across all 3 categories (favorable, intermediate and poor); Test type: Other; p < 0.0001, Log Rank
Statistical Analysis 2: Comparison: Participants With mRCC and/or aRCC: Second Line Axitinib Treatment; Data were compared statistically across all 3 categories (favorable, intermediate and poor); Test type: Other; p = 0.0004, Log Rank

6. Secondary Outcome: Overall Survival (OS): International Metastatic Renal Cell Carcinoma Database Consortium (IMDC) Stratification
Description: OS was defined as the time between the index date and the date of death from any cause. Participants who were still alive at the study end date or the last visit date available were censored. IMDC criteria had 6 risk factors: KPS <80% (ability to perform ordinary tasks, 0 [dead] -100 [normal]); time from diagnosis to start of systemic therapy <12 months; corrected serum calcium >10.0 mg/dL; neutrophils and platelets >LLN and hemoglobin <LLN. Present risk factors were added, and then participants were stratified in following prognosis group: favorable (0 factor), intermediate (1-2 factors), poor (>=3 factors), unknown/missing =no information available. Index date: date of initiation of first-line sunitinib therapy and second-line axitinib therapy.
Time Frame: as for outcome 4
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Participants With mRCC and/or aRCC: First Line Sunitinib Treatment | Participants With mRCC and/or aRCC: Second Line Axitinib Treatment
Number analyzed (Participants) | 622 | 121
Months
  Favorable: number analyzed (Participants) | 108 | 21
  Favorable | 34.103 [26.382 to 46.127] | NA [NA to NA] — Median and 95% CI was not estimable due to low number of participants with events.
  Intermediate: number analyzed (Participants) | 308 | 65
  Intermediate | 20.435 [17.150 to 23.491] | 16.394 [12.287 to 21.947]
  Poor: number analyzed (Participants) | 184 | 31
  Poor | 9.347 [7.524 to 10.842] | 8.049 [4.764 to 18.168]
  Unknown/missing (no information available): number analyzed (Participants) | 22 | 4
  Unknown/missing (no information available) | NA [NA to NA] — Median and 95% CI was not calculated as no information was available for these participants. | NA [NA to NA] — Median and 95% CI was not calculated as no information was available for these participants.
Statistical Analysis 1: Comparison: Participants With mRCC and/or aRCC: First Line Sunitinib Treatment; Data were compared statistically across all 3 categories (favorable, intermediate and poor); Test type: Other; p < 0.0001, Log Rank
Statistical Analysis 2: Comparison: Participants With mRCC and/or aRCC: Second Line Axitinib Treatment; Data were compared statistically across all 3 categories (favorable, intermediate and poor); Test type: Other; p = 0.0014, Log Rank

7. Secondary Outcome: Number of Participants With Best Overall Response (BOR) for Complete Response (CR), Partial Response (PR), Stable Disease (SD), PD and Surgical CR as Per RECIST v 1.1
Description: BOR was recorded for CR, PR, SD, PD and surgical CR. RECIST v1.1, a) CR: disappearance of target, non-target lesions and normalization of tumor markers. Pathological lymph nodes had short axis measures <10mm; b) PR: >=30% decrease in sum of measures (longest diameter for tumor lesions, short axis measure for nodes) of target lesions, taking reference baseline sum of diameters. Non-target lesions must be non-PD; c) PD: >=20% increase in sum of diameters of target lesions, taking as reference smallest sum on study, sum must demonstrate absolute increase of at least 5mm. Appearance of 1 or more new lesions; d) SD: neither shrinkage for CR/PR nor increase for PD taking as reference smallest sum of longest diameters since treatment start; e) Surgical CR: disappearance of target, non-target lesions, normalization of tumor markers, pathological lymph nodes had short axis measuring <10mm as result of surgery. Alive participants with no events were censored at final study cutoff date.
Time Frame: Start of treatment till BOR of CR, PR, PD, SD, Surgical CR, or death/initiation of new therapy, whichever occurred first; from 2002 to 30 June 2018, anytime in these 16 years (data retrieved and observed retrospectively for approximately 1.2 years)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With mRCC and/or aRCC: First Line Sunitinib Treatment | Participants With mRCC and/or aRCC: Second Line Axitinib Treatment
Number analyzed (Participants) | 622 | 121
Participants
  CR | 19 | 0
  PR | 127 | 17
  SD | 252 | 50
  PD | 145 | 33
  Surgical CR | 2 | 0
  NA/Missing (no clinical response recorded in data base) | 77 | 21

8. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants who achieved a BOR of CR or PR as per RECIST v1.1. CR was defined as disappearance of target and non-target lesions and normalization of tumor markers. Pathological lymph nodes must have short axis measures <10 mm. PR was defined as at least a 30% decrease in the sum of measures (longest diameter for tumor lesions and short axis measure for nodes) of target lesions, taking as reference baseline sum of diameters. Non-target lesions must be non-PD. PD was defined as at least a 20% increase in sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions was considered progression. Alive participants who did not have event were censored at final study cutoff date.
Time Frame: From start of treatment until CR,PR,PD,death/initiation of new therapy, whichever occurred first, from inception of database(2002) until 30 June 2018, anytime in these 16 years (from data retrieved and observed retrospectively for approximately 1.2 years)
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Participants With mRCC and/or aRCC: First Line Sunitinib Treatment | Participants With mRCC and/or aRCC: Second Line Axitinib Treatment
Number analyzed (Participants) | 622 | 121
Percentage of participants | 23.5 [20.2 to 27.0] | 14.0 [8.4 to 21.5]

9. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the time between the date of the first documented confirmed response (PR or CR) and the date of the first documented progression or death due to any cause. Alive participants who did not have event were censored at final study cutoff date. As per RECIST v1.1: CR was defined as disappearance of target and non-target lesions and normalization of tumor markers. Pathological lymph nodes short axis measures <10 mm. PR was defined as at least 30% decrease in sum of measures (tumor lesions- longest diameter and nodes- short axis) of target lesions, taking as reference baseline sum of diameters. PD was defined as at least 20% increase in sum of diameters of measured lesions taking as references smallest sum of diameters recorded on study (including baseline) and an absolute increase of >=5 mm or appearance of at least 1 new lesion.
Time Frame: From date of first documented CR/PR until PD/death/initiation of new therapy, whichever occurred first, from inception of database(2002) until 30 June 2018, anytime in these 16years (data retrieved and observed retrospectively for approximately 1.2 years)
Population: Analysis population included all eligible participants with mRCC and/or aRCC, received sunitinib as first-line treatment and/or axitinib as second-line treatment from 2002 till 30 June 2018. Required information for this outcome measure was not present in Christie NHS database. Hence, data could not be collected and analyzed for this outcome measure.
Arm/Group | Participants With mRCC and/or aRCC: First Line Sunitinib Treatment | Participants With mRCC and/or aRCC: Second Line Axitinib Treatment
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Time to Treatment Discontinuation (TTD)
Description: TTD was defined as the time between initiation of treatment to the end of treatment for any reason including PD, death, and lost-to follow up. Participants were censored on the study end date or at last office visit date without clinical or radiographic evidence of PD, whichever occurred first.
Time Frame: From start of the treatment until end of treatment, from inception of database (2002) until 30 June 2018, anytime in these 16 years (from the data retrieved and observed retrospectively for approximately 1.2 years)
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Participants With mRCC and/or aRCC: First Line Sunitinib Treatment | Participants With mRCC and/or aRCC: Second Line Axitinib Treatment
Number analyzed (Participants) | 622 | 121
Months | 8.509 [7.589 to 9.889] | 6.899 [5.158 to 9.528]

11. Secondary Outcome: Time to Treatment Discontinuation (TTD): Memorial Sloan-Kettering Cancer Center (MSKCC) Stratification
Description: TTD was defined as the time between initiation of treatment to the end of treatment for any reason including PD, death, and lost-to follow up. Participants were censored on the study end date or at last office visit date without clinical or radiographic evidence of PD, whichever occurred first. MSKCC criteria had following 5 risk factors: KPS <80% (ability to perform ordinary tasks, 0 [dead] -100 [normal]); time from diagnosis to start of systemic therapy <12 months; hemoglobin <LLN; lactate dehydrogenase 1.5*ULN; corrected serum calcium >10.0 mg/dL. Present risk factors were added, and then participants were stratified in following prognosis group: favorable (0 factor), intermediate (1-2 factors), poor (>=3 factors), unknown/missing = no information available.
Time Frame: as for outcome 10
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Participants With mRCC and/or aRCC: First Line Sunitinib Treatment | Participants With mRCC and/or aRCC: Second Line Axitinib Treatment
Number analyzed (Participants) | 622 | 121
Months
  Favorable: number analyzed (Participants) | 122 | 19
  Favorable | 15.836 [11.959 to 20.961] | 12.649 [4.895 to 16.099]
  Intermediate: number analyzed (Participants) | 378 | 72
  Intermediate | 9.051 [7.589 to 10.119] | 8.903 [5.552 to 12.222]
  Poor: number analyzed (Participants) | 85 | 17
  Poor | 2.760 [1.807 to 4.600] | 1.610 [0.690 to 2.924]
  Unknown/missing (no information available): number analyzed (Participants) | 37 | 13
  Unknown/missing (no information available) | NA [NA to NA] — Median and 95% CI was not calculated as no information was available for these participants. | NA [NA to NA] — Median and 95% CI was not calculated as no information was available for these participants.
Statistical Analysis 1: Comparison: Participants With mRCC and/or aRCC: First Line Sunitinib Treatment; Data were compared statistically across all 3 categories (favorable, intermediate and poor); Test type: Other; p < 0.0001, Log Rank
Statistical Analysis 2: Comparison: Participants With mRCC and/or aRCC: Second Line Axitinib Treatment; Data were compared statistically across all 3 categories (favorable, intermediate and poor); Test type: Other; p < 0.0001, Log Rank

12. Secondary Outcome: Time to Treatment Discontinuation (TTD): International Metastatic Renal Cell Carcinoma Database Consortium (IMDC) Stratification
Description: TTD was defined as the time between initiation of treatment to the end of treatment for any reason including PD, death, and lost-to follow up. Participants were censored on the study end date or at last office visit date without clinical or radiographic evidence of PD, whichever occurred first. IMDC criteria had following 6 risk factors: KPS <80% (ability to perform ordinary tasks, 0 [dead] -100 [normal]); time from diagnosis to start of systemic therapy <12 months; corrected serum calcium >10.0 mg/dL; neutrophils and platelets >LLN and hemoglobin <LLN. Present risk factors were added, and then participants were stratified in following prognosis group: favorable (0 factor), intermediate (1-2 factors), poor (>=3 factors), unknown/missing =no information available.
Time Frame: as for outcome 10
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Participants With mRCC and/or aRCC: First Line Sunitinib Treatment | Participants With mRCC and/or aRCC: Second Line Axitinib Treatment
Number analyzed (Participants) | 622 | 121
Months
  Favorable: number analyzed (Participants) | 108 | 21
  Favorable | 15.129 [10.809 to 20.731] | 12.649 [6.012 to 16.099]
  Intermediate: number analyzed (Participants) | 308 | 65
  Intermediate | 9.988 [8.082 to 12.189] | 7.359 [5.158 to 10.842]
  Poor: number analyzed (Participants) | 184 | 31
  Poor | 5.651 [4.830 to 6.472] | 3.680 [1.906 to 7.162]
  Unknown/missing (no information available): number analyzed (Participants) | 22 | 4
  Unknown/missing (no information available) | NA [NA to NA] — Median and 95% CI was not calculated as no information was available for these participants. | NA [NA to NA] — Median and 95% CI was not calculated as no information was available for these participants.
Statistical Analysis 1: Comparison: Participants With mRCC and/or aRCC: First Line Sunitinib Treatment; Data were compared statistically across all 3 categories (favorable, intermediate and poor); Test type: Other; p < 0.0001, Log Rank
Statistical Analysis 2: Comparison: Participants With mRCC and/or aRCC: Second Line Axitinib Treatment; Data were compared statistically across all 3 categories (favorable, intermediate and poor); Test type: Other; p = 0.0094, Log Rank

13. Secondary Outcome: Durable Response Rate (DRR)
Description: DRR was determined as the percentage of participants with objective response (CR or PR) with a duration of at least 6 months. As per RECIST v1.1: CR was defined as disappearance of target and non-target lesions and normalization of tumor markers. Pathological lymph nodes short axis measures <10 mm. PR was defined as at least 30% decrease in sum of measures (tumor lesions- longest diameter and nodes- short axis) of target lesions, taking as reference baseline sum of diameters.
Time Frame: 6 months from inception of database (2002) until 30 June 2018, anytime in these 16 years (from the data retrieved and observed retrospectively for approximately 1.2 years)
Population: as for outcome 9
Arm/Group | Participants With mRCC and/or aRCC: First Line Sunitinib Treatment | Participants With mRCC and/or aRCC: Second Line Axitinib Treatment
Number analyzed (Participants) | 0 | 0

14. Other Pre Specified Outcome: Number of Participants Who Started Systemic Therapy Within 1 Year of Diagnosis
Time Frame: Baseline (data retrieved and observed retrospectively for approximately 1.2 years)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With mRCC and/or aRCC: First Line Sunitinib Treatment | Participants With mRCC and/or aRCC: Second Line Axitinib Treatment
Number analyzed (Participants) | 622 | 121
Participants | 367 | 63

15. Other Pre Specified Outcome: Number of Participants With Karnofsky Performance Status (KPS) Less Than 80 Percent (%)
Description: KPS: used for rating participant activities of daily living on scale from 0-100, higher score = participant is better able to carry out daily activities. Score range: 100 = normal no complaints; no disease evidence, 90 = able to carry normal activity; minor signs/symptoms of disease, 80 = normal activity with effort; some signs/symptoms, 70 = cares for self; unable to carry on normal activity, 60 = requires occasional assistance, but able to care for most personal needs, 50 = requires considerable assistance and frequent medical care, 40 = disabled; requires special care, assistance, 30 = severely disabled; hospital admission is indicated although death not imminent, 20 = very sick; hospital admission necessary, 10 = moribund; fatal processes progressing rapidly and 0 = dead. The lower the score the worse is survival for most serious illnesses. Here, number of participants with KPS <80% were reported.
Time Frame: Baseline (data retrieved and observed retrospectively for approximately 1.2 years)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With mRCC and/or aRCC: First Line Sunitinib Treatment | Participants With mRCC and/or aRCC: Second Line Axitinib Treatment
Number analyzed (Participants) | 622 | 121
Participants | 89 | 28

16. Other Pre Specified Outcome: Number of Participants With Hemoglobin Less Than Lower Limit of Normal (LLN)
Description: In this outcome measure number of participants with hemoglobin less than LLN were reported. For male participants LLN was 130 grams per liter and for female participants LLN was 115 grams per liter.
Time Frame: Baseline (data retrieved and observed retrospectively for approximately 1.2 years)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With mRCC and/or aRCC: First Line Sunitinib Treatment | Participants With mRCC and/or aRCC: Second Line Axitinib Treatment
Number analyzed (Participants) | 622 | 121
Participants | 322 | 72

17. Other Pre Specified Outcome: Number of Participants With Serum Calcium >Upper Limit of Normal (ULN), Neutrophil >ULN, Platelets >ULN and Lactate Dehydrogenase >1.5*ULN
Description: Number of participants with serum calcium >ULN (3.00 millimole per liter [mmol/L]), neutrophils >ULN (7.5 *10^9/L), platelets >ULN (400 *10^9/L), lactate dehydrogenase >1.5*ULN were reported in this outcome measure.
Time Frame: Baseline (data retrieved and observed retrospectively for approximately 1.2 years)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With mRCC and/or aRCC: First Line Sunitinib Treatment | Participants With mRCC and/or aRCC: Second Line Axitinib Treatment
Number analyzed (Participants) | 622 | 121
Participants
  Serum Calcium >ULN | 45 | 7
  Neutrophil >ULN | 132 | 11
  Platelets >ULN | 181 | 28
  Lactate Dehydrogenase >1.5*ULN | 368 | 67

18. Other Pre Specified Outcome: Number of Participants Per Tumor Fuhrman Grades
Description: The four-tiered Fuhrman grading evaluates nuclear size, nuclear shape and presence of nucleolar prominence. Grade 1: small (=10 micrometer [mcm]) nuclear diameter, round/uniform nuclear shape and absent/inconspicuous nucleoli; Grade 2: large (=15 mcm) nuclear diameter, irregular outline nuclear shape and visible at *400 magnification nucleoli; Grade 3: larger (=20 mcm) nuclear diameter, obvious irregular outline nuclear shape and visible and prominent at *100 magnification nucleoli; Grade 4: grade 3 plus bizarre multilobed nuclei +/- spindle cells.
Time Frame: Baseline (data retrieved and observed retrospectively for approximately 1.2 years)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With mRCC and/or aRCC: First Line Sunitinib Treatment | Participants With mRCC and/or aRCC: Second Line Axitinib Treatment
Number analyzed (Participants) | 622 | 121
Participants
  1 | 8 | 0
  2 | 113 | 21
  3 | 141 | 34
  4 | 137 | 38
  Missing (no information available) | 223 | 28

19. Other Pre Specified Outcome: Number of Participants With Tumor Subtype
Description: In this outcome measure, number of participants were classified according to tumor subtype as clear cell, non-clear cell and unknown/missing.
Time Frame: Baseline (data retrieved and observed retrospectively for approximately 1.2 years)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With mRCC and/or aRCC: First Line Sunitinib Treatment | Participants With mRCC and/or aRCC: Second Line Axitinib Treatment
Number analyzed (Participants) | 622 | 121
Participants
  Clear cell | 484 | 102
  Non-clear cell | 54 | 7
  Unknown/missing (no information available) | 84 | 12

20. Other Pre Specified Outcome: Number of Participants With Adverse Events
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship with the study treatment.
Time Frame: From start of treatment until death, from inception of database (2002) until 30 June 2018, anytime in these 16 years (from the data retrieved and observed retrospectively for approximately 1.2 years)
Population: Minimum criteria for reporting an AE (i.e. identifiable participant, identifiable reporter, a suspect product, and event) could not met, hence, adverse events were not collected and reported.
Arm/Group | Participants With mRCC and/or aRCC: First Line Sunitinib Treatment | Participants With mRCC and/or aRCC: Second Line Axitinib Treatment
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Not applicable as adverse events were not collected during the study
Description: Minimum criteria for reporting an adverse event (i.e. identifiable participant, identifiable reporter, a suspect product, and event) could not met, hence, adverse events were not collected and reported.
Arm/Group | Participants With mRCC and/or aRCC: First Line Sunitinib Treatment | Participants With mRCC and/or aRCC: Second Line Axitinib Treatment
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Data was originally planned to be retrieved and analyzed from the database inception date (2002) until the end of June 2017. However, due to delay in data transfer, data retrieved and analysis was extended from end of June 2017 to end of June 2018. Required information for outcome measures- duration of response and durable response rate was not present in Christie NHS database. Hence, data could not be collected and analyzed for these outcome measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-14): https://cdn.clinicaltrials.gov/large-docs/91/NCT04033991/Prot_SAP_000.pdf